CLINICAL TRIAL: NCT00691769
Title: Expression of Fas Protein in Skin Biopsies of Participants With Scarring Alopecia
Status: Completed | Type: Observational
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Other Study IDs: IRB00000301; 31050
Record Dates: First submitted 2008-06-02; First posted 2008-06-05 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Central Centrifugal Scarring Alopecia; Lichen Planopilaris; Discoid Lupus Erythematosus
Keywords: alopecia; lupus
MeSH Terms: conditions — Lichen Planus; Lupus Erythematosus, Discoid; Alopecia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Two, 4mm punch biopsies will be obtained of skin tissue.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- I: CCSA subjects will be recruited from patients who have been diagnosed through biopsy with CCSA and treated with standard of care for up to eight months in the Department of Dermatology clinic of Wake Forest University School of Medicine.
- II: patients with lichen planopilaris (LP) and patients with discoid lupus erythematosus (DLE) will be collected from patients who have been diagnosed through biopsy in the clinic.
- III: Healthy study subjects will be patients from the Wake Forest University School of Medicine Department of Dermatology population undergoing excisions for cosmetic purposes or excision of free margins around tumors that would have otherwise been discarded.

SUMMARY:
The purpose of this research study is to see if a specific protein that we are interested in is involved in scarring hair loss. If these proteins are involved, further genetic work may also better define the disease as well as future treatment options.

DETAILED DESCRIPTION:
This is a single-center study, designed to evaluate the expression of Fas protein in skin biopsies of patients with scarring alopecia including fourteen patients with central centrifugal scarring alopecia (CCSA), three patients with lichen planopilaris (LP) and three patients with discoid lupus erythematosus (DLE). Skin biopsies of five healthy participants will be used as controls.

ELIGIBILITY:
Inclusion Criteria:

* Participants ages 30 years or older with a biopsy- proven diagnosis of CCSA.
* Undergone standard of care treatment for CCSA by a WFUSM Dermatologist
* Women of child bearing age will be required to have a negative pregnancy test in order to participate in the study
* Participants ages 30 years or older with a biopsy- proven diagnosis of LP.
* Participants ages 30 years or older with a biopsy- proven diagnosis of DLE.
* Healthy participants must be ages 30 years or older.

Exclusion Criteria:

* Age less than 30 years of age.
* Clinically evident bacterial or viral infection of the scalp.
* Pregnant or nursing woman of child-bearing potential.
* Participation in any other investigative research study involving study medication.
* Inability to return for the biopsy visit.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Wake Forest University Health Sciences Dermatology Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2006-04-26 (Actual); Primary Completion 2012-11-26 (Actual); Study Completion 2012-11-26 (Actual)

PRIMARY OUTCOMES:
To evaluate the expression of Fas protein in skin biopsies of participants with central centrifugal scarring alopecia (CCSA), lichen planopilaris (LP) and discoid lupus erythematosus (DLE) and in healthy controls. | 8 weeks

SECONDARY OUTCOMES:
To evaluate the expression of Fas protein in skin biopsies of participants with central centrifugal scarring alopecia before and after treatment with intralesional and topical steroids. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Amy McMichael, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences Dermatology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No